CLINICAL TRIAL: NCT04430855
Title: A Phase 2, Multicenter, Randomized, Placebo-Controlled, Double-Blind Study to Evaluate Upadacitinib in Adult Subjects With Moderate to Severe Hidradenitis Suppurativa
Brief Title: A Study of Oral Upadacitinib Tablet Compared to Placebo in Adult Participants With Moderate to Severe Hidradenitis Suppurativa to Assess Change in Disease Symptoms
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M20-040
Record Dates: First submitted 2020-06-11; First posted 2020-06-12 (Actual); Results first posted 2023-02-06 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-01

CONDITIONS: Hidradenitis Suppurativa (HS)
Keywords: Hidradenitis suppurativa (HS); Upadacitinib
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — upadacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Upadacitinib 30 mg (Experimental): Participants will receive 30 mg upadacitinib orally once a day for 12 weeks (Period 1) followed by 30 mg upadacitinib orally once a day for 36 weeks (Period 2).
  Interventions: Drug: Upadacitinib
- Placebo followed by Upadacitinib 15 mg (Experimental): Participants will receive matching placebo orally once a day for 12 weeks (Period 1) followed by 15 mg upadacitinib orally once a day for 36 weeks (Period 2).
  Interventions: Drug: Upadacitinib; Drug: Placebo

INTERVENTIONS:
Drug: Upadacitinib — Tablet; Oral
  Other Names: RINVOQ
Drug: Placebo — Tablet; Oral
  Arms: Placebo followed by Upadacitinib 15 mg

SUMMARY:
Hidradenitis suppurativa (HS) is an inflammatory skin disease that causes painful lesions in the axilla (underarm), inguinal (groin) and anogenital (anal and genital) regions. This study will evaluate how well upadacitinib compared to placebo (no medicine) works to treat hidradenitis suppurativa in adult participants with moderate to severe disease. The study will assess change in disease signs and symptoms.

DETAILED DESCRIPTION:
Upadacitinib is an investigational drug being developed for the treatment of HS. This study is "double-blinded," which means that neither the trial participants nor the study doctors will know who will be given study drug and who will receive placebo (no medicine). Participants are randomly (by chance) put into 1 of 2 groups, called treatment arms. They are randomized in a 2 to 1 ratio meaning more participants have a chance to receive upadacitinib compared to placebo.

Participants will undergo approximately 35-days of screening followed by a 48-week treatment period and a 30-day follow-up visit after the last dose of study drug for a total study duration of up to 57 weeks. The treatment period will consist of a 12-week placebo-controlled, double-blind period (Period 1) and a 36-week blinded extension period (Period 2).

There may be a higher burden for participants in this trial compared to their standard of care. Participants will attend visits every other week, once a month, or once every 2 months during the course of the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of hidradenitis suppurativa (HS) for at least 1 year prior to Baseline.
* Total abscess and inflammatory nodule (AN) count of ≥ 5 at Baseline, presence of HS lesions in at least 2 distinct anatomical areas, and draining fistula count of ≤ 20 at Baseline.
* History of inadequate response or an intolerance to adequate trial of oral antibiotics for treatment of HS.
* Required to use a daily antiseptic wash on HS lesions.

Exclusion Criteria:

-History of active skin disease (other than HS) that could interfere with assessment of HS, including skin infections requiring systemic treatment within 4 weeks of the Baseline visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2020-07-14 (Actual); Primary Completion 2021-04-22 (Actual); Study Completion 2022-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (26):
- United States (18):
  - Medical Dermatology Specialist /ID# 221084, Phoenix, Arizona
  - University of Arkansas for Medical Sciences /ID# 218404, Little Rock, Arkansas
  - Medderm Associates /ID# 218317, San Diego, California
  - Skin Care Research - Boca Raton /ID# 218809, Boca Raton, Florida
  - Lakes Research, LLC /ID# 218854, Miami, Florida
  - ForCare Clinical Research /ID# 218013, Tampa, Florida
  - Northshore University Health System Dermatology Clinical Trials Unit /ID# 218319, Skokie, Illinois
  - Dawes Fretzin, LLC /ID# 218310, Indianapolis, Indiana
  - Beth Israel Deaconess Medical Center /ID# 218306, Boston, Massachusetts
  - Washington University-School of Medicine /ID# 218331, St Louis, Missouri
  - Psoriasis Treatment Center of Central New Jersey /ID# 218330, East Windsor, New Jersey
  - Duke Cancer Center /ID# 218526, Durham, North Carolina
  - University Hospitals Case Medical Center /ID# 218326, Cleveland, Ohio
  - Southside Dermatology /ID# 218321, Tulsa, Oklahoma
  - University of Pittsburgh MC /ID# 218329, Pittsburgh, Pennsylvania
  - Medical University of South Carolina /ID# 218318, Charleston, South Carolina
  - Duplicate_Center for Clinical Studies /ID# 218307, Houston, Texas
  - Dermatology Specialists of Spokane /ID# 218760, Spokane, Washington
- Canada (4):
  - Dermatology Research Institute Inc. /ID# 218780, Calgary, Alberta
  - Winnipeg Clinic /ID# 218963, Winnipeg, Manitoba
  - Dr. Wei Jing Loo Medicine Prof /ID# 218779, London, Ontario
  - Lynderm Research Inc. /ID# 218778, Markham, Ontario
- Japan (3):
  - Takagi Dermatology Clinic /ID# 218587, Obihiro-shi, Hokkaido
  - University Hospital Kyoto Prefectural University of Medicine /ID# 220859, Kyoto, Kyoto
  - Toranomon Hospital /ID# 218588, Minato-ku, Tokyo
- Cruz-Santana, Carolina, PR /ID# 221188, Carolina, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: This clinical study may be evaluating a usage that is not currently FDA approved. Please see US Prescribing Information for approved uses. — https://www.rxabbvie.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 21 study sites in 3 countries (Canada, Japan, and United States/Puerto Rico).
Pre-assignment Details: Participants were randomized to upadacitinib or placebo in a 2:1 ratio. Randomization was stratified by anti-tumor necrosis factor (TNF) use prior to Baseline (yes or no) and Hurley stage (< III or III).
Groups:
- Placebo / Upadacitinib 15 mg: Participants received matching placebo orally once a day for 12 weeks (Period 1) followed by 15 mg upadacitinib orally once a day for 36 weeks (Period 2).
- Upadacitinib 30 mg: Participants received 30 mg upadacitinib orally once a day for 12 weeks (Period 1) followed by 30 mg upadacitinib orally once a day for 36 weeks (Period 2).
Period: Period 1 (Weeks 1-12)
Arm/Group | Placebo / Upadacitinib 15 mg | Upadacitinib 30 mg
Started | 21 | 47
Received Study Drug | 21 | 47
Completed | 19 | 41
Not Completed | 2 | 6
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Lost to Follow-up | 0 | 2
Not completed — Lack of Efficacy | 0 | 1
Not completed — Other | 0 | 1
Period: Period 2 (Weeks 12-48)
Arm/Group | Placebo / Upadacitinib 15 mg | Upadacitinib 30 mg
Started | 19 | 41
Completed | 14 | 31
Not Completed | 5 | 10
Not completed — Withdrawal by Subject | 2 | 5
Not completed — Lost to Follow-up | 1 | 2
Not completed — Lack of Efficacy | 2 | 3

BASELINE CHARACTERISTICS:
Population: The Intent-to-treat (ITT) population includes all randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo / Upadacitinib 15 mg | Upadacitinib 30 mg | Total
Number analyzed (Participants) | 21 | 47 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.6 (12.49) | 36.7 (11.70) | 36.6 (11.85)
Age, Customized [Count of Participants; unit: Participants]
  < 40 years | 15 | 29 | 44
  40 - < 65 years | 5 | 17 | 22
  ≥ 65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 37 | 53
  Male | 5 | 10 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 9 | 14
  Not Hispanic or Latino | 16 | 38 | 54
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 12 | 19
  White | 11 | 30 | 41
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Prior Exposure to Tumor Necrosis Factor (TNF) Antagonists [Count of Participants; unit: Participants]
  Yes | 6 | 12 | 18
  No | 15 | 35 | 50
Hurley Stage [Count of Participants; unit: Participants] — The Hurley staging system is a grading system to characterize the extent of disease in patients with hidradenitis suppurativa. Hurley stages are described as follows:
  * Stage I - Abscess formation, single or multiple, without sinus tracts and cicatrization (scarring)
  * Stage II - Single or multiple, widely separated, recurrent abscesses with tract formation and cicatrization
  * Stage III - Diffuse or near-diffuse involvement, or multiple interconnected tracts and abscesses across the entire area
  Participants
    Stage I | 1 | 0 | 1
    Stage II | 11 | 24 | 35
    Stage III | 9 | 23 | 32
Duration of Hidradenitis Suppurativa (HS) Disease [Mean (Standard Deviation); unit: years] | 9.83 (4.990) | 11.52 (9.401) | 11.00 (8.290)
Abscess Lesion Count [Mean (Standard Deviation); unit: abscess lesions] — Abscesses are lesions that contain fluid, are tender or painful, with or without drainage.
  abscess lesions | 4.0 (3.29) | 4.8 (6.39) | 4.6 (5.60)
Inflammatory Nodule Lesion Count [Mean (Standard Deviation); unit: nodule lesions] — Tender, small lumps under the skin that are inflamed or reddened,
  nodule lesions | 15.7 (12.77) | 18.4 (20.98) | 17.6 (18.78)
Draining Fistula Lesion Count [Mean (Standard Deviation); unit: draining fistula lesions] — Horizontal channels (or tunnels) below the skin that connect the lesions and open into a sore on the skin surface that releases fluid (pus).
  draining fistula lesions | 4.3 (6.17) | 3.4 (4.74) | 3.7 (5.19)
Abscess and Inflammatory Nodule (AN) Count [Mean (Standard Deviation); unit: abscesses and inflammatory nodules] | 19.8 (12.87) | 23.2 (24.64) | 22.1 (21.65)
Patient's Global Assessment (PGA) of Skin Pain Score [Mean (Standard Deviation); unit: units on a scale] — Participants were asked to rate their worst skin pain in the last 24 hours on an 11-point numerical rating scale (NRS) ranging from 0 (no skin pain) to 10 (skin pain as bad as you can imagine) on a daily basis using an electronic diary.
  Baseline PGA skin pain score is defined as the last non-missing weekly average score, calculated based on the daily scores from the past 7 days (with non-missing values in 4 or more days of the 7 day period), before the date of the first administration of study drug. Population: Participants with available data
  units on a scale
    number analyzed (Participants) | 20 | 45 | 65
    (all) | 4.852 (3.3237) | 4.987 (2.7120) | 4.945 (2.8879)
PGA Skin Pain Score In Participants with a Baseline Value ≥ 3 [Mean (Standard Deviation); unit: units on a scale] — Participants were asked to rate their worst skin pain in the last 24 hours on an 11-point numerical rating scale ranging from 0 (no skin pain) to 10 (skin pain as bad as you can imagine) on a daily basis using an electronic diary.
  Baseline PGA skin pain score is defined as the last non-missing weekly average score, calculated based on the daily scores from the past 7 days (with non-missing values in 4 or more days of the 7 day period), before the date of the first administration of study drug. Population: Participants with a Baseline PGA skin pain score ≥ 3
  units on a scale
    number analyzed (Participants) | 12 | 33 | 45
    (all) | 7.168 (2.0395) | 6.180 (2.1107) | 6.444 (2.1155)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Hidradenitis Suppurativa Clinical Response (HiSCR) at Week 12
Description: HiSCR is defined as at least a 50% reduction in the total abscess and inflammatory nodule (AN) count with no increase in abscess count and no increase in draining fistula count relative to Baseline.
Time Frame: Baseline and Week 12
Population: Intent-to-treat population; participants with missing data at Week 12 due to a missing assessment or early discontinuation, for reasons other than coronavirus disease 2019 (COVID-19), and participants who initiated antibiotics for HS-related infections prior to Week 12 were counted as non-responders (non-responder imputation); missing data due to COVID-19 infection or logistical restriction were handled by multiple imputation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Placebo: Participants received matching placebo orally once a day for 12 weeks.
- Upadacitinib 30 mg: Participants received 30 mg upadacitinib orally once a day for 12 weeks.
Arm/Group | Placebo | Upadacitinib 30 mg
Number analyzed (Participants) | 21 | 47
percentage of participants | 23.8 [5.6 to 42.0] | 38.3 [24.4 to 52.2]
Statistical Analysis 1: Comparison: Upadacitinib 30 mg; The primary analysis compared the percentage of participants in the upadacitinib 30 mg treatment group who achieved HiSCR response to that of a prespecified, single historical placebo rate (25%). The historical placebo rate of 25% was assumed based on the corresponding response rates of placebo participants satisfying the same key eligibility criteria from the 2 adalimumab HS Phase 3 studies, Study M11-313 (NCT01468207) and Study M11-810 (NCT01468233); Test type: Superiority; p = 0.018, Chi-squared; Response Rate Difference = 13.3, 95% CI 2-sided [-0.6 to 27.2] — Response rate difference compared to historical placebo = upadacitinib 30 mg - historical placebo
Statistical Analysis 2: Comparison: Upadacitinib 30 mg; As a supplemental analysis, the percentage of participants who achieved HiSCR at Week 12 was further analyzed by comparing upadacitinib with in-trial placebo participants combined with subjects with historical placebo HiSCR data pre-selected using propensity score matching from adalimumab studies M11-313 and M11-810 and risankizumab study M16-833 (NCT03926169), whose study populations, entry criteria and study designs were similar to this study. The placebo in-trial + synthetic HiSCR was 29.2%; Test type: Superiority; p = 0.142, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline Hurley Stage [Stage < III, Stage III] and prior TNF use [Yes or No]); Adjusted Response Rate Difference = 9.2, 95% CI 2-sided [-7.6 to 25.9] — Response rate difference = upadacitinib 30 mg - placebo (in-trial + synthetic)
Statistical Analysis 3: Comparison: Placebo vs Upadacitinib 30 mg; As an additional supplemental analysis, the percentage of participants who achieved HiSCR at Week 12 was also analyzed by comparing upadacitinib 30 mg with in-trial placebo participants; Test type: Superiority; p = 0.087, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 2]; Adjusted Response Rate Difference = 14.7, 95% CI 2-sided [-6.6 to 36.0] — Response rate difference = upadacitinib 30 mg - placebo

2. Secondary Outcome: Percentage of Participants Achieving PGA Skin Pain Numeric Rating Scale 30 (NRS30) Response at Week 12 Among Participants With Baseline NRS ≥ 3
Description: The Patient's Global Assessment (PGA) of Skin Pain Numeric Rating Scale (NRS) was used to assess the worst skin pain due to HS. Participants were asked to rate their worst skin pain in the last 24 hours on an 11-point numerical rating scale ranging from 0 (no skin pain) to 10 (skin pain as bad as you can imagine) on a daily basis using an electronic diary. The weekly average score was calculated based on the daily scores from the 7 days prior to the visit (with non-missing values in 4 or more days of the 7 day period).
  NRS30 is defined as the percentage of participants who achieved at least a 30% reduction and at least 1 unit reduction from Baseline in the PGA of skin pain NRS in participants with Baseline skin pain NRS ≥ 3.
Time Frame: Baseline and Week 12
Population: Intent-to-treat population with Baseline skin pain NRS ≥ 3; participants with missing data at Week 12 due to a missing assessment or early discontinuation, for reasons other than COVID-19, and participants who initiated antibiotics for HS-related infections prior to Week 12 and under the impact of analgesic use at Week 12 were counted as non-responders (non-responder imputation); missing data due to COVID-19 infection or logistical restriction were handled by multiple imputation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 30 mg
Number analyzed (Participants) | 12 | 33
percentage of participants | 33.3 [6.7 to 60.0] | 36.4 [20.0 to 52.8]
Statistical Analysis 1: Comparison: Upadacitinib 30 mg; The primary analysis compared the percentage of participants in the upadacitinib 30 mg treatment group who achieved NRS30 response to that of a prespecified, single historical placebo rate (22.5%). The historical placebo rate of 22.5% was assumed based on the corresponding response rates of placebo participants satisfying the same key eligibility criteria from the 2 adalimumab HS Phase 3 studies, Study M11-313 (NCT01468207) and Study M11-810 (NCT01468233); Test type: Superiority; p = 0.028, Chi-squared; Response Rate Difference = 13.9, 95% CI 2-sided [-2.5 to 30.3] — Response rate difference compared to historical placebo (upadacitinib 30 mg - historical placebo)
Statistical Analysis 2: Comparison: Upadacitinib 30 mg; As a supplemental analysis, the percentage of participants who achieved NRS30 at Week 12 was further analyzed by comparing upadacitinib with in-trial placebo participants combined with subjects with historical placebo NRS30 data pre-selected using propensity score matching from adalimumab studies M11-313 and M11-810 and risankizumab study M16-833 (NCT03926169), whose study populations, entry criteria and study designs were similar to this study. The placebo in-trial + synthetic NRS30 was 31.3%; Test type: Superiority; p = 0.323, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel test adjusted for strata (Baseline Hurley Stage [Stage < III, Stage III] and prior TNF use [Yes or No]); Adjusted Response Rate Difference = 4.5, 95% CI 2-sided [-14.6 to 23.5] — Response rate difference = upadacitinib 30 mg - placebo (in-trial + synthetic)
Statistical Analysis 3: Comparison: Placebo vs Upadacitinib 30 mg; As an additional supplemental analysis, the percentage of participants who achieved NRS30 at Week 12 was also analyzed by comparing upadacitinib 30 mg with in-trial placebo participants; Test type: Superiority; p = 0.421, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 2]; Adjusted Response Rate Difference = 2.2, 95% CI 2-sided [-19.6 to 24.0] — Response rate difference = upadacitinib 30 mg - placebo

ADVERSE EVENTS:
Time Frame: Period 1: From first dose of study drug up to the first dose of study drug during Period 2 (12 weeks). Period 2: From first dose of study drug in Period 2 up to 30 days after the last dose of study drug (maximum of 40 weeks).
Groups:
- Period 1: Placebo: Participants received matching placebo orally once a day for 12 weeks in Period 1.
- Period 1: Upadacitinib 30 mg: Participants received 30 mg upadacitinib orally once a day for 12 weeks in Period 1.
- Period 2: Upadacitinib 15 mg: Participants originally assigned to placebo received 15 mg upadacitinib orally once a day for 36 weeks in Period 2.
- Period 2: Upadacitinib 30 mg: Participants originally assigned to upadacitinib 30 mg continued to receive 30 mg upadacitinib orally once a day for 36 weeks in Period 2.
Arm/Group | Period 1: Placebo | Period 1: Upadacitinib 30 mg | Period 2: Upadacitinib 15 mg | Period 2: Upadacitinib 30 mg
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/47 | 0/19 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/21 | 3/47 | 0/19 | 5/41
Other Adverse Events (participants affected / at risk) | 6/21 | 12/47 | 10/19 | 12/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Period 1: Placebo (N=21) | Period 1: Upadacitinib 30 mg (N=47) | Period 2: Upadacitinib 15 mg (N=19) | Period 2: Upadacitinib 30 mg (N=41)
CHOLECYSTITIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CELLULITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ADJUSTMENT DISORDER (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DEPRESSION (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SUICIDAL BEHAVIOUR (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SUICIDAL IDEATION (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HIDRADENITIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SKIN PLAQUE (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ABORTION INDUCED (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPOTENSION (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Period 1: Placebo (N=21) | Period 1: Upadacitinib 30 mg (N=47) | Period 2: Upadacitinib 15 mg (N=19) | Period 2: Upadacitinib 30 mg (N=41)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CHILLS (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FATIGUE (General disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
MALAISE (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
PYREXIA (General disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
BRONCHITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CELLULITIS (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 3 (4) | 0 (0) | 2 (2)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
DIZZINESS (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
HEADACHE (Nervous system disorders) | 0 (0) | 5 (5) | 2 (2) | 2 (2)
ABNORMAL DREAMS (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ACNE (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 3 (4)
DERMATITIS (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
ECZEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HIDRADENITIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (4) | 3 (3)
PERIORAL DERMATITIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PRURITUS ALLERGIC (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2020-10-25): https://cdn.clinicaltrials.gov/large-docs/55/NCT04430855/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-30): https://cdn.clinicaltrials.gov/large-docs/55/NCT04430855/SAP_001.pdf